CLINICAL TRIAL: NCT03268525
Title: The Effect of Local Anesthesia on Postoperative Pain in Vaginal Hysterectomy: A Randomized Controlled Trial
Brief Title: The Effect of Local Anesthesia on Postoperative Pain in Vaginal Hysterectomy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Ohad Gluck, OBGYN resident, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 0156-17-WOMC
Record Dates: First submitted 2017-08-22; First posted 2017-08-31 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Drug group versus placebo group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The surgeons, the pain assessing researchers, and the participating women will all be blinded to what the syringes contain.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study (Active Comparator): Marcaine 0.5 % Injectable Solution will be injected before incision, and in a systematic fashion as a modified paracervical block. First, 2 ml will be injected through the vaginal fornices at 03.00, 06.00, 09.00, and 12.00 hours at 2 cm depth. Thus, 8 ml will be systematically injected around the cervical circumference before incision. In addition, 1 ml of the solution will be injected in each resection line (sacro-uterine and cardinal ligaments), adding up to a total of 10 ml. In case of performing additional anterior/ posterior colporrhaphy, additional solution of Marcaine 0.25%will be prepared: 5 ml of the solution will be injected to the cutting line of the anterior/ posterior vaginal wall, respectively, prior to incision.
  Interventions: Drug: Marcaine 0.5 % Injectable Solution
- Control (Placebo Comparator): Sodium Chloride 0.9% will be injected before incision, and in a systematic fashion as a modified paracervical block. First, 2 ml will be injected through the vaginal fornices at 03.00, 06.00, 09.00, and 12.00 hours at 2 cm depth. Thus, 8 ml will be systematically injected around the cervical circumference before incision. In addition, 1 ml of the solution will be injected in each resection line (sacro-uterine and cardinal ligaments), adding up to a total of 10 ml. In case of performing additional anterior/ posterior colporrhaphy, additional solution of Sodium Chloride 0.9% will be prepared: 5 ml of the solution will be injected to the cutting line of the anterior/ posterior vaginal wall, respectively, prior to incision.
  Interventions: Drug: Sodium Chloride 0.9%

INTERVENTIONS:
Drug: Marcaine 0.5 % Injectable Solution — Local infiltration by Marcaine 0.5% Injectable Solution prior to incision
  Other Names: Study
  Arms: Study
Drug: Sodium Chloride 0.9% — Local infiltration by Sodium Chloride 0.9% prior to incision
  Other Names: Placebo
  Arms: Control

SUMMARY:
The investigators aim is to study the effect of pre-operative local anesthetic on post vaginal hysterectomy pain.

DETAILED DESCRIPTION:
This is a double-blinded, randomized, controlled trial. Women who undergone elective vaginal hysterectomy and gave their informed consent were included. Exclusion criteria included additional abdominal, chronic pelvic pain, malignancy, and allergy to Bupivacaine.

Solutions of either Bupivacaine-Hydrochloride 0.5%, or Sodium-Chloride 0.9% as a placebo, were prepared prior to surgery, according to randomization. The chosen solution was injected before incision, as a modified paracervical block, and in each resection line (sacro-uterine and cardinal ligaments). The amount of fluid administered was 10 ml. When colporrhaphy was also performed, an additional 5 ml of solution were injected in the midline of the vaginal wall prior to each incision line.

By utilizing the 10 cm Visual-analogue-scale (VAS) we examined the differences in post-operative pain at rest at 3, 8, and 24 hours, and during ambulation at 8 and 24 hours using multivariate linear regression models. We also assessed the differences in analgesics given at the different time points between the groups using multivariate negative binomial regression models.

ELIGIBILITY:
Inclusion Criteria:

* Elective vaginal hysterectomy on benign indication

Exclusion Criteria:

additional abdominal, chronic pelvic pain, malignancy, and allergy to Bupivacaine.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Pain at movement | 24 hours
  Movement-evoked pain will be scored after the operation

SECONDARY OUTCOMES:
pain at rest | 24 hours
  Pain at rest will be scored with the woman lying in bed after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Shimon Ginat, MD, Study Director — Wolfson Medical Center
Locations (1):
- Wolfson medical center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No